CLINICAL TRIAL: NCT01781377
Title: Randomized Controlled Trial of Prophylactic Subhypnotic Propofol vs Metoclopramide and in Combination Therapy for the Prevention of Nausea and Vomiting During Subarachnoid Anesthesia for Cesarean Section.
Brief Title: Prophylactic Subhypnotic Propofol for Nausea and Vomiting During for Cesarean Section Under Subarachnoid Anesthesia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Collaborators: Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Zhirajr Mokini, M.D., Azienda Ospedaliera San Gerardo di Monza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1632/08 COET
Record Dates: First submitted 2013-01-25; First posted 2013-02-01 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: PREGNANCY
Keywords: NAUSEA; VOMITING; CESAREAN SECTION; PREVENTION; PROPOFOL
MeSH Terms: conditions — Nausea; Vomiting | interventions — Propofol; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PROPOFOL (Experimental): PROPOFOL SINGLE BOLUS 10 mg + 1mg/kg/hr INFUSION AT UMBILICAL CORD RESECTION
  Interventions: Drug: PROPOFOL
- METOCLOPRAMIDE (Experimental): METOCLOPRAMIDE 10 mg I.V. AT UMBILICAL CORD RESECTION
  Interventions: Drug: METOCLOPRAMIDE
- PROPOFOL & METOCLOPRAMIDE (Experimental): PROPOFOL SINGLE BOLUS of 10 mg + 1mg/kg/hr INFUSION AND METOCLOPRAMIDE 10 mg I.V. AT UMBILICAL CORD RESECTION
  Interventions: Drug: PROPOFOL; Drug: METOCLOPRAMIDE
- PLACEBO (Placebo Comparator): SALINE INFUSION
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: PROPOFOL — PROPOFOL FOR NAUSEA AND VOMITING PROPHYLAXIS
  Arms: PROPOFOL; PROPOFOL & METOCLOPRAMIDE
Drug: METOCLOPRAMIDE — METOCLOPRAMIDE FOR NAUSEA AND VOMITING PROPHYLAXIS
  Arms: METOCLOPRAMIDE; PROPOFOL & METOCLOPRAMIDE
Drug: PLACEBO — SALINE INFUSION
  Arms: PLACEBO

SUMMARY:
Perioperative nausea and vomiting may occur in 50-80% of patients undergoing cesarean section.

Metoclopramide is a well known Dopamine receptor antagonist that acts at the Chemoreceptor trigger zone and is used effectively for the prevention and treatment of nausea and vomiting. Propofol can antagonize Serotonin receptors in the area postremal and is associated to a reduced incidence of postoperative nausea and vomiting. Some studies have shown that propofol can prevent intraoperative nausea and vomiting during cesarean section.

The control of risk factors and the pharmacological prophylaxis of nausea and vomiting reduces effectively their incidence.

In this randomized, double blind, case-control study the efficacy of propofol alone, metoclopramide alone and in combination in controlling nausea and vomiting were compared. A risk factor control strategy was associated to each study group.

ELIGIBILITY:
Inclusion Criteria:

CESAREAN SECTION WITHOUT MATERNAL OR FETAL SUFFERING

American Society of Anesthesiologists score I-II

36 TO 41 WEEK OF GESTATION

BMI < 35

HEMOGLOBIN > 10 mg/dl

NO COMPLICATIONS (GESTATIONAL DIABETES, COLESTASIS)

NO ACUTE OR CHRONIC GASTROINTESTINAL DISORDERS (GERD excluded)

NO SMOKING OR DRUG ABUSE DURING PREGNANCY

NO PREVIOUS MAJOR ABDOMINAL SURGERY

NO PREVIOUS COMPLICATED PREGNANCIES

FETAL WEIGHT > 2.5 kg

Exclusion Criteria:

EMERGENCY CESAREAN SECTION WITH MATERNAL OR FETAL SUFFERING

American Society of Anesthesiologists score III-IV-V

< 36 OR > 41 WEEK OF GESTATION

BMI > 35

HEMOGLOBIN < 10 mg/dl

COMPLICATIONS (GESTATIONAL DIABETES, COLESTASIS)

ACUTE OR CHRONIC GASTROINTESTINAL DISORDERS

SMOKING OR DRUG ABUSE DURING PREGNANCY

PREVIOUS MAJOR ABDOMINAL SURGERY

PREVIOUS COMPLICATED PREGNANCIES

FETAL WEIGHT < 2.5 kg

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2008-02; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
NAUSEA AND VOMITING ASSOCIATED WITH CESAREAN SECTION | FROM ANESTHESIA TO THE END OF SURGERY (AVERAGE 2 HOURS)
  INCIDENCE OF NAUSEA AND VOMITING

SECONDARY OUTCOMES:
ADVERSE EVENTS | FROM ANESTHESIA TO THE END OF SURGERY (AVERAGE 2 HOURS)
  HEADACHE, AGITATION, SEDATION.

CONTACTS AND LOCATIONS:
Overall Officials: ZHIRAJR MOKINI, M.D., Principal Investigator — Azienda Ospedaliera San Gerardo di Monza; FLAVIA PETRINI, M.D., Study Director — University of Chieti; MICHELE SCESI, M.D., Study Director — University of Chieti
Locations (1):
- A.O. SS.ma Annunziata, Chieti, Italy, Italy